CLINICAL TRIAL: NCT06268015
Title: Botensilimab and Balstilimab Optimization in Colorectal Cancer (BBOpCo)
Brief Title: Botensilimab and Balstilimab Optimization in Colorectal Cancer
Acronym: BBOpCo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nicholas DeVito, MD (Other)
Collaborators: Gateway for Cancer Research (Other); Agenus Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nicholas DeVito, MD, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115311
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: metastatic; unresectable; microsatellite stable; MSS; untreated; first-line; 1st line
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — balstilimab; Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): botensilimab + balstilimab until disease progression, then botensilimab + balstilimab + mFOLFOX6 (leucovorin, fluorouracil, oxaliplatin) + {bevacizumab or panitumumab}
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Bevacizumab; Drug: Panitumumab

INTERVENTIONS:
Drug: Botensilimab — 75 mg IV every 6 weeks for up to 4 doses
Drug: Balstilimab — 240 mg IV every 2 weeks
Drug: Oxaliplatin — 85 mg/m2 IV every 2 weeks
Drug: Leucovorin — 400 mg/m2 IV every 2 weeks
Drug: Fluorouracil — 400 mg/m2 IV bolus + 2,400 mg/m2 IV (over 46 hours) every 2 weeks
Drug: Bevacizumab — 5 mg/kg IV every 2 weeks
Drug: Panitumumab — 6 mg/kg IV every 2 weeks

SUMMARY:
This is a single-arm, interventional, pilot clinical trial. Fifteen evaluable patients will have tumor-informed ctDNA testing at baseline and start botensilimab and balstilimab treatment. They will receive botensilimab and balstilimab in 6-week cycles until progression, after which mFOLFOX6 and bevacizumab or panitumumab will be added to the regimen. Subjects will have safety testing at baseline and every two weeks while on study drug. Study treatment with botensilimab and balstilimab, mFOLFOX6, and bevacizumab or panitumumab will be continued until radiographic or clinical progression, toxicity, or patient withdrawal. Subjects will have one safety follow up visit 30 days after the last treatment and will be followed for survival every 12 weeks for up to 2 years.

DETAILED DESCRIPTION:
3.1 Study Description

This is a single-arm, interventional, pilot clinical trial. Subjects with newly diagnosed, metastatic or unresectable, microsatellite stable colorectal cancer without liver, bone, or brain metastases will start study treatment with botensilimab and balstilimab alone. They will have restaging scans every 6 weeks. When the subject experiences progression on the study drug(s), they may choose to add mFOLFOX6 and either bevacizumab or panitumumab to the combination. The determinant of whether the subject crosses over will be radiographic progression (iCPD) per iRECIST. Subjects will continue on the new combination until radiographic or clinical progression, intolerable toxicity, or patient withdrawal.

No more than 20 subjects will be enrolled to ensure the trial obtains 15 evaluable subjects. All patients will be enrolled at the Duke Cancer Institute.

* Enrolled subjects are defined as subjects who give informed consent.
* Screen failures are defined as subjects who give informed consent and do not meet eligibility criteria.
* Accrued subjects are defined as subjects who give informed consent and meet eligibility criteria.

  * Withdrawal: Subject accrued but later withdrawn from the study, either before or after receiving a study drug.
  * Evaluable: All subjects who are accrued and receive any infusion from Cycle 1 study treatment with botensilimab and balstilimab will be evaluable for safety. Subjects who are accrued, receive C1 study treatment, and complete the first cycle of safety assessments will be considered evaluable for the primary endpoints of disease control rate and safety.
  * Non-evaluable: Subjects who accrued but did not complete the first cycle of safety assessments due to reasons other than study treatment-attributed toxicity (e.g., disease progression or inter-current illness) are considered non-evaluable for safety and efficacy.

Study Treatment Botensilimab 75 mg IV Every 6 weeks for up to 4 doses Balstilimab 240 mg IV Every 2 weeks Oxaliplatin 85 mg/m2 IV Every 2 weeks Leucovorin 400 mg/m2 IV Every 2 weeks Fluorouracil 400 mg/m2 IV bolus Every 2 weeks Fluorouracil 2400 mg/m2 IV Every 2 weeks (over 46 hours) Bevacizumab 5 mg/kg IV Every 2 weeks Panitumumab 6 mg/kg IV Every 2 weeks

3.2 Crossover Criteria

Patients are treated with first line botensilimab and balstilimab with plans to add chemotherapy if they experience iCPD per iRECIST. Once the subject has iRECIST confirmed progression, they can add SOC therapy as described in section 3.1. Subject must meet the following criteria to qualify for treatment beyond progression on ICB therapy:

* Absence of signs or symptoms indicating clinically significant PD
* No decline in ECOG performance status
* Absence of any of the investigational product discontinuation criteria
* Lead PI approval

The decision to discontinue botensilimab and balstilimab at any point prior to or during the addition of chemotherapy will be made by the PI or patient or if a clinically significant Grade 4 AE occurs.

5.1 Screening Period

During the Screening Period, subjects are consented and screened for the study. Informed consent must be obtained before initiation of any screening procedure that is performed solely for the purpose of determining eligibility for this study. Evaluations performed as part of routine care before informed consent can be considered as screening evaluations if done within the defined screening period, and if permitted by the local Institutional Review Board (IRB)/ Independent Ethics Committee (IEC) policies. Study eligibility is based on meeting all of the inclusion criteria and none of the exclusion criteria before the first dose of study drug on Cycle 1 Day 1.

The following study procedures must be done within 28 days prior to Cycle 1 Day 1:

* Inclusion and exclusion criteria
* Demographics
* Medical and cancer history
* Physical examination
* Height
* Vital signs and weight
* Concomitant medications
* CT and/or MRI of chest, abdomen, and pelvis
* PT/INR (prior to fresh tissue biopsy)
* Fresh tissue biopsy
* Archived tissue collection

The following study procedures must be done or repeated within 7 days prior to Cycle 1 Day 1:

* CBC with differential
* CMP
* TSH and fT4
* Pregnancy test (only for people of childbearing potential)

Subject eligibility is determined using lab results obtained up to 7 days prior to Cycle 1 Day 1. Any laboratory assessments repeated on Cycle 1 Day 1 must meet eligibility requirements. The Screening Period ends upon receipt of the first dose of study drug or final determination that the subject is ineligible for the study.

5.2 Treatment Period

During the Treatment Period, subjects will receive botensilimab every 6 weeks for up to 4 doses and balstilimab every 2 weeks for up to 2 years. Following progression on the study drug(s), mFOLFOX6 will be administered every 2 weeks. Investigators will choose between bevacizumab and panitumumab, which will be administered every 2 weeks. Cycle length is every 6 weeks, with study visits occurring every 2 weeks. A treatment window of ± 2 days is allowed for day 1 of cycle 2 and all subsequent cycles. The Treatment Period lasts until: 1) subject has been receiving balstilimab for 2 years; 2) disease progression; 3) the occurrence of unacceptable treatment-attributed toxicity; or 4) other reason(s) for subject discontinuation as described in Section 5.7. Toxicity-attributed dose modifications of any of the study drugs may occur during the Treatment Period.

After the completion of the first cycle, laboratory assessments may be obtained up to 2 days prior to treatment. If necessary, the treatment visit may be within ± 2 days of the scheduled day 1 for cycle 2 and all subsequent cycles. If clinically indicated, additional visits and/or safety assessments may be warranted.

The following study procedures must be completed on days 1, 15, and 29 of each cycle:

* Concomitant medications
* Physical examination
* Vital signs and weight
* ECOG performance status
* CBC with differential
* CMP
* Pregnancy test (only for people of childbearing potential)
* Administer balstilimab
* Administer mFOLFOX6 (if applicable)
* Administer bevacizumab (if applicable)
* Administer panitumumab (if applicable)
* Adverse event assessment

The following study procedures must be added to the above test/procedures prior to dosing on Day 1 of each cycle:

* Plasma for ctDNA
* Plasma for CEA
* Administer botensilimab (maximum 4 doses)

Blood for biomarker analysis will be collected prior to treatment on C1D1 and C3D1 only.

Restaging scans and tumor assessment (CT and/or MRI scans) will be performed every 6 weeks while on study drug(s) alone, then every 8 weeks after crossover (±1 week). Disease response will be assessed using the guidelines described in Section 5.6.

Thyroid function tests (TSH and fT4) must be completed every 12 weeks (every other cycle; i.e., baseline, C3, C5, C7, etc)

The following study procedures must be completed at time of progression on study drug(s) (any time prior to the start of chemotherapy administration):

* Optional biopsy of the progressing lesion
* PT/INR (only if doing biopsy, prior to biospy)
* Plasma for ctDNA
* Plasma for CEA
* Blood for biomarker analysis

The Treatment Period ends when a subject receives his or her last dose of study treatment; the subject then enters the Follow-up Period.

5.3 Follow-up Period

Subjects should return 30 (±7) days after their last dose of study drug for an end-of-treatment visit to complete the following study procedures:

* Concomitant medications
* Physical examination
* Vital signs and weight
* ECOG performance status
* Adverse event assessment
* CBC with differential
* CMP
* Thyroid profile (TSH and fT4)
* Serum pregnancy test (only for people of childbearing potential)
* Plasma for ctDNA
* Plasma CEA
* Blood for biomarker analysis

Subjects will have a telephone visit with the study team at 90 (±7) days after the last dose of study drug to complete an AE assessment. Any delayed irAEs must be reported to the PI.

Subjects with adverse events (AEs) attributed to study drug that are ongoing at the time of this 90-day safety follow-up visit will continue to be followed unless the AE is deemed unresolvable or the subject has started a new anti-cancer treatment regimen.

For subjects that are discontinued from study treatment for reasons other than disease progression, subjects will have disease status (blood tumor marker(s) and restaging scans per standard of care schedule) followed until disease progression or start of new anti-cancer treatment regimen. Disease status may be collected via personal interviews or review of medical records.

Subjects will be followed for survival up to 2 years after discontinuing the study drug regimen or until the study is closed (whichever comes first). Survival status may be collected by phone call or review of medical or public records every 12 (±2) weeks.

5.4 Laboratory Assessments

Local laboratories will perform all clinical laboratory tests using standard procedures, and results will be provided to the Investigator. Abnormalities in clinical laboratory tests that lead to a change in subject management (e.g., dose modification, requirement for additional medication, treatment or monitoring) are considered clinically significant for the purposes of this study and will be recorded on the case report form (CRF). If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as a serious adverse event (SAE). Refer to Appendix D for details of laboratory tests for this study.

5.5 Adverse Event Assessment

AEs will be documented throughout the study. AE seriousness, grade, and relationship to study drug will be assessed by the investigator using NCI-CTCAE version 5.0.

5.6 Tumor Assessments

Tumor response will be assessed using RECIST v.1.1 and iRECIST. Radiographic imaging will be performed with CT scan of chest/abdomen/pelvis with and without contrast and/or MRI scan of abdomen/pelvis every 6 weeks while on botensilimab and balstilimab alone, then every 8 weeks after crossover. The same method for tumor assessment should be employed at every assessment.

If a subject has unconfirmed progressive disease (iUPD) per iRECIST, they may continue on study until they have confirmed progressive disease (iCPD) provided that they meet all of the following criteria:

1. No deterioration in ECOG performance status
2. Clinical benefit from continued treatment, per investigator assessment
3. Patient is tolerating study drug
4. Patient has no clinical symptoms indicating clear disease progression
5. Continued treatment will not prevent or delay treatment that would otherwise prevent serious complications of their disease.

5.7 Subject Discontinuation

Subjects will receive study treatment until treatment discontinuation for one of the reasons listed below. However, subjects may discontinue study treatment or withdraw their consent to participate in the study at any time without prejudice. All reasons for discontinuation or withdrawal from trial will be recorded.

Subjects who progress on the initial study drug regimen do not have to discontinue study treatment at that time. Rather, they will add mFOLFOX6 and either bevacizumab or panitumumab and continue on study treatment. Patients who have complete response or prolonged stable disease may also elect to end study therapy after a discussion with their treating physician and with approval of the PI. Reasons for subject discontinuation may include, but are not limited to, the following:

* Subject has been receiving balstilimab for 2 years
* Occurrence of any clinically significant grade 4 AE
* Death
* Confirmed radiographic disease progression after switching to the botensilimab and balstilimab plus chemo/bev/pmab
* Significant noncompliance by subject or Investigator
* Investigator or Lead PI determination that it is no longer safe and/or no longer in the subject's best interest to continue participation
* Withdrawal of consent
* Loss to follow-up
* Necessity for treatment with other anticancer treatment prohibited by protocol
* Sexually active subjects who refuse to follow the contraceptive guidelines
* Women who become pregnant or are breast feeding
* Request by regulatory agencies for termination of treatment of an individual subject or all subjects under the protocol
* Discontinuation of treatment may be considered for participants who have attained a confirmed complete response (iCR).

ELIGIBILITY:
Inclusion Criteria:

1. Participants of any gender who are at least 18 years of age on the day of signing informed consent.
2. Histologically confirmed metastatic and/or unresectable colorectal cancer without liver metastasis or known or suspected bone or brain metastases.

   a. Subjects with lung, lymph node, and locoregional sites of disease (primary tumor or serosal implant) are permitted. Patients with peritoneal carcinomatosis may be included unless they have clinically relevant ascites (See exclusion 17).
3. Microsatellite stable disease, as documented in the participant's medical record at the time of consent by the absence of MSI-H or dMMR result in an FDA-approved assay or an IVD offered as an LDT that includes microsatellite stability biomarker.
4. Subject must be willing to provide fresh biopsy of tumor lesion. *Note: Those who do not have a tumor lesion that is safe and amenable to biopsy may still be enrolled.
5. ECOG performance status of 0 or 1.
6. No prior systemic therapy for colon cancer.

   a. Subjects who received systemic therapy in the neoadjuvant or adjuvant setting completed at least 6 months prior to enrollment are eligible.
7. Measurable disease per RECIST v1.1.
8. People of child-bearing potential must not be pregnant or breast feeding and meet at least one of the following conditions:

   1. Not a person of childbearing potential (POCBP)
   2. A POCBP must agree to use a reliable method of contraception (refer to Section 6.7.1) during the treatment period and for at least 180 days after the last dose of study treatment.
9. All participants must practice effective contraceptive methods (refer to section 6.7.1) during the treatment period, unless documentation of infertility exists.
10. Expected to survive >3 months per investigator assessment.
11. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
12. Adequate organ function as defined below. Specimens must have been collected within 7 days prior to the start of study treatment:

    * Absolute neutrophil count (ANC) ≥1,500/µL
    * Platelets ≥100,000/µL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the last 2 weeks)
    * Measured or calculated creatinine clearance (GFR can be used in place of CrCl) ≥45 mL/min (Creatinine clearance (CrCl) should be calculated per institutional standard)
    * Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels > 1.5 x ULN
    * AST (SGOT) and ALT (SGPT) ≤2.5 x ULN
    * International normalized ratio (INR) OR prothrombin time (PT) ≤1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Prior therapy with an immune checkpoint inhibitor.
2. A POCBP who is pregnant or breastfeeding or has a positive pregnancy test within 72 hours prior to receiving study treatment
3. Not willing to use an effective method of birth control as defined in section 6.7.1
4. Known liver, bone, or CNS metastases and/or carcinomatous meningitis.
5. Diagnosis of other carcinomas within the last 2 years, except cured non-melanoma skin cancer, treated thyroid cancer, curatively treated in-situ cervical cancer, or localized prostate cancer treated curatively with no evidence of biochemical or imaging recurrence.
6. Documented history of clinically significant autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, type 1 diabetes mellitus, psoriasis not requiring systemic treatment, well-controlled hypothyroidism, or conditions not expected to recur in the absence of and external trigger are permitted to enroll.
7. Any history of chronic or autoimmune pancreatitis.
8. Known history of or any evidence of active, non-infectious pneumonitis.
9. Current use of medications specified by the protocol as prohibited for administration in combination with study drug.

   1. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to the start of study drug are not eligible.
   2. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
   3. Corticosteroids administered as pre-medication for IV contrast allergy are also allowed.
10. Received a live vaccine within 30 days prior to the start of study drug.

    1. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. However, intranasal influenza vaccines (e.g. Flu-Mist) are live-attenuated vaccines, and are not allowed within 28 days of study treatment
    2. COVID-19 vaccines will be allowed. However, COVID vaccines are not allowed within 7 days of starting study drug treatment
11. Recent or current active infectious disease requiring systemic antivirals, antibiotics or antifungals, or treatment within 2 weeks prior to the start of study drug.
12. Concurrent severe and/or uncontrolled medical conditions, which may compromise participation in the study, including impaired heart function or clinically significant heart disease.
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the start of study drug (56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study.
14. Serious, non-healing wound, ulcer, or bone fracture.
15. Patients with a history of organ or allogenic hematopoietic stem cell transplantation.
16. Partial or complete bowel obstruction within the last 3 months, signs/ symptoms of bowel obstruction, or known radiologic evidence of impeding obstruction.
17. Refractory ascites defined as requiring 2 or more therapeutic paracenteses within the last 4 weeks or ≥4 times within the last 90 days or ≥1 time within the last 2 weeks prior to study entry or requiring diuretics within 2 weeks of study entry.
18. Tumor location or size that may result in life-threatening complications. For example, lesions that may put patient at risk for intestinal perforation or obstruction.
19. Known or suspected allergy or hypersensitivity to any investigational or standard of care therapy agents, or any of the inactive ingredients in any of the components of the study drug regimen.
20. Peripheral neuropathy from prior neoadjuvant or adjuvant oxaliplatin must have resolved to G2 or lower.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Disease control rate based on iRECIST at second restaging scan | 24 weeks after screening
  Disease control rate is defined as the proportion of subjects who have a complete response, partial response, or stable disease at the time of a second restaging scan. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease is defined as a decrease of less than 30% or an increase of less than 20%. Increases of 20% or greater must be confirmed 4-8 weeks later, and confirmation scans must also show an increase of at least 5 mm in the sum of lesion sizes or an increase in the number of lesions. Otherwise, the increase will be counted as stable disease.
Proportion of subjects with a best overall response of complete response or partial response according to iRECIST | up to 2 years
  The number of subjects who went on treatment and had a complete response or partial response sometime during the study (prior to progression) divided by the number of subjects who went on treatment.

SECONDARY OUTCOMES:
Disease control rate based on RECIST v1.1 at second restaging scan | 24 weeks after screening
  Disease control rate is defined as the proportion of subjects who have a complete response, partial response, or stable disease at the time of a second restaging scan. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease is defined as a decrease of less than 30% or an increase of less than 20%.
Proportion of subjects with a best overall response of complete response or partial response according to RECIST v1.1 | up to 2 years
  The number of subjects who went on treatment and had a complete response or partial response sometime during the study (prior to progression) divided by the number of subjects who went on treatment.
Months of overall survival | up to 2 years
  Months from treatment start date until the date of death from any cause.
Months of progression-free survival | up to 2 years
  Months from treatment start date until the date of first documented radiographic progression or date of death from any cause (whichever is first). Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No